CLINICAL TRIAL: NCT01704482
Title: N-acetylcysteine for Renal Protection in Patients With Rheumatic Heart Disease Undergoing Valve Replacement.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Samy Abbas, assistant lecturer of anesthesia and ICU, Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: tafanono01003060187
Record Dates: First submitted 2012-10-09; First posted 2012-10-11 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Cardiac Surgery for Rheumatic Valvular Heart Disease; Renal Dysfunction
MeSH Terms: conditions — Renal Insufficiency | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- N-acetylcysteine (Experimental): N-acetylcysteine bolus of 150 mg/kg in 250 mL of 5% glucose over 15 mins, followed by continuous intravenous infusion of 50 mg/kg in 250 mL of 5% glucose over 4 hrs, then 100 mg/kg in 1000 ml of 5% glucose over 20 hrs
  Interventions: Drug: N-acetylcysteine
- Glucose 5% (Placebo Comparator): equivalent volume over the same period.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: N-acetylcysteine — NAC bolus of 150 mg/kg in 250 mL of 5% glucose over 15 mins, followed by continuous intravenous infusion of 50 mg/kg in 250 mL of 5% glucose over 4 hrs, then 100 mg/kg in 1000 ml of 5% glucose over 20 hrs
  Arms: N-acetylcysteine
Drug: placebo
  Arms: Glucose 5%

SUMMARY:
We aim to investigate the efficacy of N-acetylcysteine (NAC) to attenuate acute renal dysfunction in patients with rheumatic valvular heart disease undergoing single valve replacement.

ELIGIBILITY:
Inclusion Criteria:

* patients with rheumatic heart disease undergoing single valve replacement

Exclusion Criteria:

* End stage renal disease (plasma creatinine concentration ≥ 300 µmol/L)
* Emergency cardiac surgery
* Planned off-pump cardiac surgery
* Chronic inflammatory disease on immunosuppression
* Chronic moderate to high dose corticosteroid therapy (≥ 10 mg/day prednisone or equivalent)
* Age ≤ 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Absolute change in serum creatinine from baseline to peak level | within 5 days after surgery

SECONDARY OUTCOMES:
the relative change in serum creatinine. | the first five postoperative days

OTHER OUTCOMES:
the urinary output | the first five postoperative days

CONTACTS AND LOCATIONS:
Overall Officials: Laila H Mohamed, Prof, Study Chair — Assiut university hosiptal; Nawal A Gad El-rab, Prof, Study Director — Assiut university hosiptal; Fatma A Abd El-Aal, Ass Prof, Study Director — Assiut university hosiptal
Locations (1):
- Assiut University hospital, Asyut, Egypt